CLINICAL TRIAL: NCT04800692
Title: The Effects of ATLAS (Arginine Tetrahydrobiopterin L-Ascorbate) Therapy on Nitric Oxide Bioavailability and Pain-free Walking in Patients With Intermittent Claudication
Brief Title: The Effects of ATLAS Therapy on Nitric Oxide Bioavailability in Patients With Intermittent Claudication
Acronym: ATLAS
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Louis Messina (Other)
Collaborators: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor-Investigator, Louis Messina, Professor, University of Massachusetts, Worcester
Organization: University of Massachusetts, Worcester (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: H00012734
Record Dates: First submitted 2021-03-11; First posted 2021-03-16 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Claudication, Intermittent; Peripheral Artery Disease; Peripheral Vascular Diseases
MeSH Terms: conditions — Intermittent Claudication; Peripheral Arterial Disease; Peripheral Vascular Diseases | interventions — sapropterin; Arginine

STUDY DESIGN:
Intervention Model Description: All subjects will receive the same starting dose of the 3 components which will be escalated at day 45.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Tetrahydrobiopterin Dose 1 (Day 0 to 44) (Experimental): All subjects will receive 3300mg l-Ascorbate , l-Arginine 3400mg and 10mg/kg of Tetrahydrobiopterin once a day.
  Interventions: Drug: Tetrahydrobiopterin 10 mg/kg; Drug: L-Ascorbate; Drug: L-Arginine
- Tetrahydrobiopterin Dose 2 (Day 45 to 90) (Experimental): All subjects will receive 3300mg l-Ascorbate, l-Arginine 3400mg and 20mg/kg of Tetrahydrobiopterin once a day.
  Interventions: Drug: Tetrahydrobiopterin 20 mg/kg; Drug: L-Ascorbate; Drug: L-Arginine

INTERVENTIONS:
Drug: Tetrahydrobiopterin 10 mg/kg — 10mg/kg of Tetrahydrobiopterin daily.
  Other Names: sapropterin; kuvan
  Arms: Tetrahydrobiopterin Dose 1 (Day 0 to 44)
Drug: Tetrahydrobiopterin 20 mg/kg — 20mg/kg of Tetrahydrobiopterin daily.
  Other Names: sapropterin; kuvan
  Arms: Tetrahydrobiopterin Dose 2 (Day 45 to 90)
Drug: L-Ascorbate — 3300 mg of l-ascorbate once daily
Drug: L-Arginine — 3400mg of l-arginine once daily

SUMMARY:
This study will focus on people with claudication from peripheral arterial disease. The investigators are researching whether a multicomponent therapeutic can increase the production of Nitric Oxide in the blood and whether that leads to an improvement in pain free walking distance and overall physical activity.

DETAILED DESCRIPTION:
The primary objective of this study is to show that ATLAS Therapy, (L-Arginine; Tetrahydrobiopterin; L-Ascorbate) is bioavailable in humans and exerts a measurable effect on its in vivo biological signature, Flow Mediated Vasodilation (FMD) in people with intermittent claudication caused by peripheral arterial disease. This will be a Phase I / dose finding study. All subjects will receive 2 different drug doses of the Kuvan the first 45 days they will receive 10 mg/kg/day. The second 45 days they will receive 20/mg/kg/day.

ELIGIBILITY:
Inclusion Criteria:

* PAD as demonstrated by an ABI <0 .9 in one leg or TBI less than <0.7 in patients with an ABI >1.3 (non compressible vessels)
* Rutherford Classification II, III
* Age >18 years old
* Willingness to discontinue phosphodiesterase (PDE) 5 inhibitors such as Viagra, Cialis, Levitra, Revatio
* Willingness to discontinue phosphodiesterase (PDE) 3inhibitors cilostazol, milrinone or Vesnarinone
* Willing and able to comply with all study procedures
* Willing and able to provide informed consent
* Sexually active subjects willing to use an acceptable method of contraception while participating in the study

Exclusion Criteria:

* Hypotension defined as a systolic blood pressure less than 100mmhg systolic at screening or baseline visit
* Critical Leg Ischemia (Rutherford Classification IV, V, VI)
* Surgical intervention to alleviate symptoms of claudication in the study leg within the past 6 months or any endovascular interventions within 3 months or who is scheduled to undergo surgical revascularization in the next 6 month
* Walking limited by reasons other than claudication (e.g. arthritis, lung disease, severe neuropathy, lower extremity amputation except single digits)
* Serum creatinine >1.5mg/dl or Hepatic enzymes >2X the upper limit of normal
* Serum potassium greater than 5.0 or use of a potassium sparing diuretic at screening
* Pregnant, breast feeding or planning to become pregnant (subject or partner) at any time during the study.
* Myocardial Infarction, Cerebrovascular Accident or deep vein thrombosis within 12 months of screening
* Known history of nephrolithiasis
* History of ever having a seizure
* Concurrent disease or condition that would interfere with study participation or safety such as bleeding disorders, organ transplant, long term immunosuppression (excluding inhaled steroids), current neoplasm or severe gastroesophageal reflux
* History of vertigo or syncope within the past 10 years
* Enrollment in another drug or device study within 30 days of screening
* Required treatment with a drug known to inhibit folate metabolism (e.g. Methotrexate)
* Taking any of the following medications; PDE3 Inhibitors, PDE5 inhibitors, trental, nitrates, ginkgo biloba, levodopa, warfarin,
* Axillary lymph node dissection
* Presence of an amputation except single digits in either leg
* Preexisting illness that limits ambulation such as severe COPD, class III-IV heart failure, severe arthritis or back pain
* Glucose-6-dehydrogenase deficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-06-15 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Nitric Oxide bioavailability | 90 days
  Nitric Oxide bioavailability as measured by flow mediated dilatation (FMD).

CONTACTS AND LOCATIONS:
Overall Officials: Louis M Messina, MD, Principal Investigator — UMASS Medical School
Locations (1):
- UMASS Memorial Healthcare - University Campus, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No